CLINICAL TRIAL: NCT03746210
Title: Non-Invasive Characterization of Focal Liver Lesions in Liver Cirrhosis
Acronym: NICETIES
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Michael Praktiknjo, Principal Investigator / Medical Doctor, University Hospital, Bonn
Other Study IDs: NICETIES
Record Dates: First submitted 2018-11-14; First posted 2018-11-19 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Liver Cirrhoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Standard diagnostic procedures — B-Mode ultrasound, Duplex sonography, contrast-enhanced ultrasound, elastography, CT, MRI, anthropometrics

SUMMARY:
This study aims to analyze non-invasive characterization focal liver lesions in patients with liver cirrhosis. The diagnostic accuracy and predictive value of non-invasive methods is studied.

DETAILED DESCRIPTION:
This study aims to analyze non-invasive characterization focal liver lesions in patients with liver cirrhosis. The diagnostic accuracy and predictive value of non-invasive methods is studied.

Upon diagnosis multiparametric ultrasound imaging of the lesions as well as sarcopenia parameters are performed for characterization of the lesions. For primary endpoint the results are then analyzed with regard to diagnostic accuracy compared to gold standard (CT, MRI or histology). For secondary endpoint, predictive value of the non-invasive diagnostics are analyzed with regards to mortality and response to treatment.

All work up, treatment and follow up are applied in standard of care fashion.

ELIGIBILITY:
Inclusion Criteria:

* all patients with focal liver lesions and liver cirrhosis

Exclusion Criteria:

* no consent
* under 18 years

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes all adult patients in our institution with liver cirrhosis and diagnosis of focal liver lesions. Non-invasive charaterization (multiparametric ultrasound, sarcopenia assessment) and standard of care work up, treatment and follow up is applied to all patients.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | 1 year
  The diagnostic accuracy of non-invasive imaging of focal liver lesions in liver cirrhosis compared to gold standard (histology, CT and/or MRI)

SECONDARY OUTCOMES:
Predictive Value | up to 5 years
  The predictive value on mortality and treatment response of non-invasive imaging of focal liver lesions in liver cirrhosis

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: Undecided